CLINICAL TRIAL: NCT06557603
Title: Single Dose Bioequivalence Study of Ivermectin 1% Cream and Soolantra (Ivermectin) 10 mg/g Cream in Healthy Adult Human Subjects
Brief Title: Bioequivalence Study of Ivermectin 1% Cream and Soolantra (Ivermectin) 10 mg/g Cream
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Humanis Saglık Anonim Sirketi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: C1B01784
Record Dates: First submitted 2024-08-14; First posted 2024-08-16 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Rosacea
MeSH Terms: conditions — Rosacea | interventions — Ivermectin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ivermectin cream (Experimental): Ivermectin 1% cream
  Interventions: Drug: Ivermectin cream; Drug: Soolantra ® (Ivermectin) cream
- Soolantra (Ivermectin) cream (Active Comparator): Soolantra (Ivermectin) 10 mg/g cream
  Interventions: Drug: Ivermectin cream; Drug: Soolantra ® (Ivermectin) cream

INTERVENTIONS:
Drug: Ivermectin cream — [1 gm ± 0.030 gm] of product was applied in a thin layer over the entire face (avoiding the eyes, lips, and mucous membranes).
Drug: Soolantra ® (Ivermectin) cream — [1 gm ± 0.030 gm] of product was applied in a thin layer over the entire face (avoiding the eyes, lips, and mucous membranes).

SUMMARY:
Single dose bioequivalence study of Ivermectin 1% cream and Soolantra (Ivermectin) 10 mg/g cream in healthy adult human subjects.

DETAILED DESCRIPTION:
An open label, randomized, four-period, two treatment, two-sequence, fully replicate, crossover, balanced, single dose bioequivalence study.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 45 years old, both inclusive.
* Gender: Male and/or non-pregnant, non-lactating female. A. Female of childbearing potential had a negative serum beta human chorionic gonadotropin (β-HCG) pregnancy test performed within 28 days prior to first cream application day. They has used an acceptable form of contraception.

B. For female of childbearing potential, acceptable forms of contraception included the following:

i. Non hormonal intrauterine device in place for at least 3 months prior to the start of the study and remaining in place during the study period, or ii. Barrier methods containing or used in conjunction with a spermicidal agent, or iii. Surgical sterilization or iv. Practicing sexual abstinence throughout the course of the study.

C. Female was not considered of childbearing potential if one of the following was reported and documented on the medical history:

i. Postmenopausal with spontaneous amenorrhea for at least one year, or ii. Bilateral oophorectomy with or without a hysterectomy and an absence of bleeding for at least 6 months, or iii. Total hysterectomy and an absence of bleeding for at least 3 months.

* BMI: 18.5 to 30.0 kg/m2, both inclusive; BMI value were rounded off to one significant digit after decimal point (e.g. 30.04 rounded down to 30.0, while 18.45 rounded up to 18.5).
* Volunteer having weight ≥ 50 Kg.
* The Volunteers were able to communicate effectively with study personnel.
* The Volunteers willing to provide written informed consent to participate in the study.
* All volunteers were judged by the principal or sub-investigator or physician as normal and healthy during a pre-study safety assessment performed within 28 days of the first dose of cream application which included:

  1. A physical examination (clinical examination) with no clinically significant finding.

Exclusion Criteria:

Volunteers who met any one of the following criteria were not enrolled in the study.

* History of allergic responses to Ivermectin or other related drugs, or any of its formulation ingredients.
* Female subjects of childbearing potential had unprotected sexual intercourse with any non-sterile male partner (i.e. male who was not sterilized by vasectomy for at least 6 months) within 14 days prior to the first dose of cream application.
* Currently pregnant, lactating or breast-feeding (for female volunteers).
* Use of oral contraceptives within 30 days prior to the first dose of cream application (for female volunteers).
* Had significant diseases or clinically significant abnormal findings during screening [medical history, physical examination (clinical examination), laboratory evaluations, ECG recording, gynecological history and examination (including pelvic examination and routine breast examination) (for female volunteers)].
* Any disease or condition like diabetes, psychosis or others, which compromised the haemopoietic, gastrointestinal, renal, hepatic, cardiovascular, respiratory, central nervous system or any other body system.
* History or presence of bronchial asthma.
* Use of any hormone replacement therapy within 3 months prior to the first dose of cream application.
* A depot injection or implant of any drug within 3 months prior to the first dose of cream application.
* Use of CYP enzyme inhibitors or inducers within 30 days prior to the first dose of cream application.
* History or evidence of drug dependence or of alcoholism or of moderate alcohol use.
* Smokers who smoked 10 or more cigarettes per day or 20 or more biddies per day or those who could not refrained from smoking during the study period.
* History of difficulty with donating blood or difficulty in accessibility of veins.
* A positive hepatitis screen (includes subtypes B & C).
* A positive test result for HIV antibody.
* Volunteers who had received a known investigational drug within seven elimination half life of the administered drug prior to the first dose of cream application.
* Volunteers who had donated blood or loss of blood 50 ml to 100 ml within 30 days or 101 ml to 200 ml within 60 days or >200 ml within 90 days (excluding volume drawn at screening for this study) prior to first dose of cream application, whichever was greater.
* Sitting systolic blood pressure less than 100 mmHg or greater than 140 mmHg or sitting diastolic blood pressure less than 60 mmHg or greater than 90 mmHg and pulse rate less than 60 or greater than 100 beats per minute during screening.
* Illness within 14 days before the start of the study.
* Hospitalisation within 3 months before the start of the study (at the discretion of the Investigator).
* Intolerance to venipuncture.
* Any food allergy, intolerance, restriction or special diet that, in the opinion of the principal investigator or sub-investigator, contraindicated the volunteer's participation in this study.
* Institutionalized volunteers.
* Use of any prescribed medications within 14 days prior to the first dose of cream application.
* Use of any OTC products, vitamin and herbal products, etc., within 7 days prior to the first dose of cream application.
* Use of grapefruit and grapefruit containing products within 7 days prior to the first dose of cream application.
* Ingestion of any caffeine or xanthine products (i.e. coffee, tea, chocolate, and caffeinecontaining sodas, colas, etc.), cigarettes and tobacco containing products, recreational drugs, alcohol or other alcohol containing products within 48 hours prior to the first dose of cream application.
* Ingestion of any unusual diet, for whatever reason (e.g.: low sodium) for three weeks prior to the first dose of cream application.
* Volunteer has tattoo, mark of injury/surgery, any discolouration of skin, any ongoing skin disease or history of frequent skin disease, damaged skin at application sites or has cracks/hardening/scarring at the application site.
* Presence of open sores, or other skin abnormalities at the application site.
* History of cryodestruction or chemodestruction, dermabrasion, photodynamic therapy, intralesional steroids within one month.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — 36 Male + 08 Female
Enrollment: 44 (Actual)
Dates: Start 2024-03-06 (Actual); Primary Completion 2024-07-11 (Actual); Study Completion 2024-07-22 (Actual)

PRIMARY OUTCOMES:
Maximum measured plasma concentration (Cmax) | 21 hours
  If the reference product intra-subject CV is less than or equal to 30% for Cmax, then the 90% confidence interval of the relative mean Cmax of the test to reference formulation for Ln-transformed data was to be within 80.00% to 125.00%.
Area under the plasma concentration versus time curve from the time zero time point to the last quantifiable concentration (AUCt) | 21 hours
  The 90% confidence interval of the relative mean (Geometric mean) of the Test to reference formulation for Ln-transformed AUCt was to be within 80.00% to 125.00%

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve from time zero to infinity (AUCi) | 21 hours
  Descriptive statistic
Time of the maximum measured plasma concentration (Tmax) | 21 hours
  Descriptive statistic

CONTACTS AND LOCATIONS:
Locations (1):
- Cliantha Research Limited, Vadodara, Gujarat, India

IPD SHARING:
Plan to Share IPD: No